CLINICAL TRIAL: NCT00717275
Title: A Phase II Study of Temozolomide (TMZ) Following Stereotactic Radiosurgery (SRS) for Patients With Newly Diagnosed Brain Metastases
Brief Title: Study of Temozolomide to Treat Newly Diagnosed Brain Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: METS-001
Record Dates: First submitted 2008-07-15; First posted 2008-07-17 (Estimated); Results first posted 2012-07-12 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-07

CONDITIONS: Brain Metastases
Keywords: Brain Metastases; Temozolomide; Temodar; TMZ; Stereotactic Radiosurgery; SRS
MeSH Terms: conditions — Brain Neoplasms | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Temozolomide (Experimental)
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — 75 mg/m2 taken by mouth once a day for 14 out of 28 consecutive days until progression or unacceptable toxicity.
  Other Names: Temodar; TMZ

SUMMARY:
The purpose of this study is to determine if administering temozolomide after completion of stereotactic radiosurgery helps control existing brain metastases and prevents the developement of new brain metastases.

DETAILED DESCRIPTION:
Brain metastases represent a heterogenous group of system tumors whose presence in the central nervous system result in profound neurological devastation. Existing therapies for brain metastases are focused on improving both neurologic function and survival. Therapies aimed at controlling the tumor both at the site of the brain metastases and the rest of the brain have the potential to improve outcomes and quality of life. The combined use of stereotactic radiosurgery followed by temozolomide may represent such a strategy.

ELIGIBILITY:
Inclusion Criteria:

Tumor characteristics adequate for stereotactic radiosurgery:

1. 1-3 newly diagnosed, previously untreated, brain metastases
2. Each tumor measuring a size less than or equal to 3 cm
3. No other contraindications to stereotactic radiosurgery

Systemic parameters adequate for temozolomide following stereotactic radiosurgery:

1. Histological confirmation of systemic malignancy (brain confirmation not required)
2. Male or female 18 years of age or older
3. Negative pregnancy test (if of childbearing potential)
4. Any number of previous recurrences will be allowed
5. Karnofsky Performance Status > 60
6. Hematocrit > 30,000
7. White blood cell count > 1,500
8. Platelet > 100,000
9. Absolute Neutrophil Count > 1,000
10. Bilirubin < 1.5 x upper limits of normal
11. Transaminases (ALT and AST) < 1.5 x upper limits of normal
12. Creatinine < 1.5 x upper limits of normal
13. Adequate medical health to participate in this study
14. Adequate documentation of menopause (natural/surgical) or patient commitment to routine use of reliable birth control (barrier/hormonal)
15. Ability to read and understand the informed consent document
16. Ability and willingness to follow all requirements of the study including following all directions, taking medication as prescribed and completing all diaries and forms
17. No other contraindications to temozolomide (severe organ dysfunction, immunosuppression, etc.)
18. Medical stability and/or recovery from effects of stereotactic radiosurgery

Exclusion Criteria:

1. Karnofsky Performance Status < 60
2. Hematocrit < 30,000
3. White blood cell count < 1,500
4. Platelet < 100,000
5. Absolute Neutrophil Count < 1,000
6. Bilirubin >1.5 x upper limits of normal
7. Transaminases (ALT and AST) > 1.5 x upper limits of normal
8. Creatinine > 1.5 x upper limits of normal
9. Inability to undergo gadolinium-contrasted MRIs, including severe claustrophobia or insufficient allergy prophylaxis
10. Germ cell, leukemia, and lymphoma histologies will be excluded
11. Prior chemotherapy or radiotherapy for brain metastases (prior resection and steroids are allowed)
12. Contraindications to radiosurgery or temozolomide chemotherapy
13. Uncontrolled systemic malignancy
14. Chemotherapy or other systemic therapy for systemic malignancy within a specified time of temozolomide initiation, depending on half-life of agent:

    1. Cytotoxic chemotherapy within the previous 4 weeks
    2. Nitrosurea (CCNU, BCNU) within the previous 6 weeks
    3. Gliadel or temozolomide within the previous 4 weeks
    4. Bevacizumab or other antiangiogenic agent within the previous 4 weeks
    5. Other targeted molecular or antibody agent within the previous 4 weeks
    6. Hormonal agent within the previous 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-09; Primary Completion 2011-01 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin M Dunbar, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the investigator's clinical practice between September 2008 and January 2011.
Groups:
- Temozolomide: Temozolomide 75mg/m2 taken by mouth on days 1-21 out of a 28 day month.
Period: Overall Study
Arm/Group | Temozolomide
Started | 3
Completed | 0
Not Completed | 3
Not completed — Premature study termination. | 3

BASELINE CHARACTERISTICS:
Arm/Group | Temozolomide
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Developed Distant Brain Failure at One Year.
Time Frame: 1 Year
Population: Data was not analyzed.
Arm/Group | Temozolomide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event monitoring began after the first dose of temozolomide and continued until study termination.
Arm/Group | Temozolomide
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide (N=3)
ALT (Metabolism and nutrition disorders) | 2 (2)
AST (Metabolism and nutrition disorders) | 2 (2)
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (1)
Bladder infection (Renal and urinary disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Insomnia (General disorders) | 1 (1)
Muscloskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Swollen lymph node (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This single center study was terminated early due to slow accrual; therefore, statistical analysis of the 3 participants was not done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes